CLINICAL TRIAL: NCT06296446
Title: Assessment of Functioning and Disability of People With Fibrimyalgia in Poland
Brief Title: Disability of People With Fibromyalgia in Poland
Status: Recruiting | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Agnieszka Sozanska, dr hab. n. o zdr., prof. UR, University of Rzeszow
Other Study IDs: disability fibromyalgia
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia; Disabilities Multiple
Keywords: fibromyalgia; disability evaluation; functioning; WHODAS 2.0; FIQ; BDI
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- people with fibromyalgia: People with fibromyalgia in Poland. The study does not include any intervention. The collected data, in a cross-sectional study, are intended to assess the functioning and disability of people with fibromyalgia using standardized questionnaires such as: WHODAS 2.0, FIQ, BDI.

SUMMARY:
Fibromyalgia is a syndrome characterized by chronic, generalized pain in muscles and joints with the presence of characteristic, symmetrically occurring so-called "tender points" - areas of the body that are excessively sensitive to pressure. The condition is associated with a feeling of chronic fatigue, mood and sleep disturbances and a sensation of body stiffness. These complaints are bothersome and significantly impair patients' functioning in every aspect of their lives. There are few studies evaluating the functioning and disability of people with fibromyalgia. No such study has been conducted in Poland to date. Therefore, the purpose of this study is to evaluate the functioning and disability of fibromyalgia patients and the relationship of the level of disability with selected factors, such as pain intensity, emotional state, sleep quality, etc.

DETAILED DESCRIPTION:
Fibromyalgia is a disease syndrome characterized by chronic, generalized muscle and joint pain with characteristic, symmetrical so-called tender points, i.e. places of the body excessively sensitive to pressure. This disease is associated with the feeling of chronic fatigue, mood and sleep disorders, and the feeling of body stiffness. These ailments are troublesome and significantly worsen the functioning of patients in every aspect of their lives. There is little research examining functioning and disability in people with fibromyalgia. No such study has been conducted in Poland so far. Therefore, the aim of the study is to assess the functioning and disability of people suffering from fibromyalgia and the relationship between the level of disability and selected factors, such as: pain intensity, emotional state, sleep quality, etc.

The study will be conducted among people suffering from fibromyalgia and associated with the National Association of Fibromyalgia Patients FIBRO-MY. The study will be conducted using an online survey created in a "Google form". The survey will include such research tools as: WHODAS 2.0 disability assessment questionnaire, Fibromyalgia Impact Questionnaire FIQ, Beck Depression Inventory BDI. The study will be conducted based on the International Classification of Functioning Disability and Health. Appropriate statistical models will be selected to analyze the data and the results will be presented in a descriptive form.

Description of research tools:

1. The WHO Disability Assessment Schedule (WHODAS 2.0) 36-item is used to measure general disability and disability in six domains: Do1 Cognition (6 items), Do2 Mobility (5 items), Do3 Self-care (4 items), Do4 Getting along (5 items), Do5 Life activities (8 items), and Do6 Participation (8 items). During the interview, the response refers to the last 30 days. Answers to the questions are rated on a 5-point scale identifying the level of di culty or problem (1 = none; 2 = mild; 3 = moderate; 4 = severe; 5 = extreme or cannot to do). The obtained results are converted according to the instructions on the scale from 0 to 100. When assessing the level of disability with the WHODAS 2.0, the following scale (consistent with the ICF) was used: no disability or an insufficient problem (0-4%), mild disability or a small problem (5-24%), moderate disability or a significant problem (25-49%), severe disability or a big problem (50-95%), and extreme disability or a total problem (96-100%).
2. The Fibromyalgia Impact Questionnaire (FIQ) The FIQ questionnaire allows us to assess the impact of fibromyalgia on the quality of life of patients. The reminder period for FIQ is 1 week. FIQ consists of 20 items examining 10 subscales (scoring dimensions): Physical functioning, Well-being, Work related, Do work, Pain, Fatigue, Rested, Stiffness, Anxiety, Depression. Individual domains are scored according to the conversion key. Once the initial scoring is complete, the scores obtained are converted to normalized scores from 0 to 10, with 0 meaning no impairment and 10 meaning maximum impairment. The total score is expressed on a scale of 0-100. Higher scores mean a greater (negative) impact of the disease on the patient's quality of life.
3. The Beck's Depression Inventory (BDI) The BDI contains 21 items on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms). The reminder period for BDI is 2 weeks. Anxiety symptoms are not assessed, but affective, cognitive, somatic, and vegetative symptoms are considered, reflecting the Diagnostic and Statistical Manual (DSM-IV) criteria for major depression. The minimum score is 0 and the maximum score is 63. Higher scores indicate greater severity of symptoms. In non-clinical populations, scores above 20 indicate depression. In people diagnosed with depression, scores of 0-13 indicate minimal depression, 14-19 (mild depression), 20-28 (moderate depression) and 29-63 (severe depression).

At least 700 people are planned to be included in the study. The study will cover people belonging to the National Association of Fibromyalgia Patients FIBRO-MY. These will be adults diagnosed with fibromyalgia who give informed consent to participate in the study and decide to complete the electronic survey. Since the study will be conducted based on an anonymous online survey, at the beginning of the study there will be information about expressing informed consent to participate in the study and a note that completing the survey is a confirmation of consent.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 and over
* People suffering from fibromyalgia
* People who give informed consent to participate in the study

Exclusion Criteria:

Tłumaczenie

* Underage persons
* People without fibromyalgia
* People who do not give informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with fibromyalgia in Poland.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
disability | 2024-01/2024-05
  Disability assessment using the WHO Disability Assessment Schedule. (WHODAS 2.0). The obtained results are converted on the scale from 0 to 100. When assessing the level of disability with the WHODAS 2.0, the following scale (consistent with the ICF) was used: no disability or an insufficient problem (0-4%), mild disability or a small problem (5-24%), moderate disability or a significant problem (25-49%), severe disability or a big problem (50-95%), and extreme disability or a total problem (96-100%).

SECONDARY OUTCOMES:
functioning | 2024-01/2024-05
  Functioning assessment using The Fibromyalgia Impact Questionnaire (FIQ). The total score is expressed on a scale of 0-100. Higher scores mean a greater (negative) impact of the disease on the patient's quality of life.
depression | 2024-01/2024-05
  Depression assessment using Beck's Depression Inventory (BDI). Scores of 0-13 indicate minimal depression, 14-19 (mild depression), 20-28 (moderate depression) and 29-63 (severe depression).
Sociodemographic data | 2024-01/2024-05
  eg. age, sex, education level, work status, number of comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Sozańska, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszow, Rzeszów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No